# **Informed Consent**

2021-1-18

Study Title: Application of Visual Laryngeal Mask Airway Combined with Endotracheal

Intubation in Non-head and Neck Surgery Under General Anesthesia

Investigator: Xia Ruan Tel: 86-13691512741

Affiliation: Peking Union Medical College Hospital

## 1. Study Objectives:

- 1) Compare the intubation time, intubation times and intubation success rate of endotracheal intubation through laryngeal mask airway under visual and non-visual conditions.
- 2) Compare the displacement rate of laryngeal mask airway after endotracheal intubation removal under visual and non-visual conditions.
- 3) Compare the incidence of oropharyngeal pain and hoarseness after endotracheal intubation through laryngeal mask airway under visual and non-visual conditions.

### 2. Study content, methods, and procedures:

After you enter this study, the anesthesiologist will ask you and collect your basic information and preoperative data, including measuring vital signs and signing the conversation, then you will be randomly divided into visual intubation group or non-visual intubation group. During the operation, your vital signs, medication, ventilation, recovery, and other indicators will be recorded. At the end of the operation, the anesthesiologist will follow you up before leaving the recovery room and the first day after the operation to record your oropharynx pain, hoarseness, nausea, vomiting and so on.

#### 3. Possible risks and benefits of participation in the study:

The anesthetic techniques and monitoring methods used in this project are all routine anesthetic techniques approved by our country, so it will not increase the risk of surgery and anesthesia.

- 1) Possible risks: patients with gastroesophageal reflux or satiety may have aspiration when using laryngeal mask airway, so such patients need to be excluded from this study. The incidence of oropharyngeal pain caused by laryngeal mask is significantly lower than that of tracheal intubation. However, some patients still have oropharyngeal discomfort, and generally it will be recovered within two to three days after operation; the rest of the risk is the same as conventional endotracheal intubation general anesthesia.
- 2) Possible benefits: 1) Visual laryngeal mask placement and visual guidance endotracheal intubation can improve the accuracy of laryngeal mask alignment, reduce the number of times to adjust the laryngeal mask position, and improve the success rate of endotracheal intubation; 2) Laryngeal mask has less airway stimulation, so removing endotracheal tube and keeping laryngeal mask to maintain mechanical ventilation can reduce or even completely avoid coughing during recovery.
- 4. Consultation on the relevant content: You have the right to consult about the content of the study, your rights, or the associated risks. You can call 86-10-69152001 for consultation at any time.

- 5. Withdrawal from the study: Your participation in this study is entirely voluntary. If for any reason, you are unwilling to participate or unwilling to continue to participate in this study, there will be no impact on your rights and treatment. In addition, you can withdraw from this study at any time, for any reason and without any loss. If you don't follow your doctor's instructions, or if your doctor considers your health and benefits, the doctor or investigator may also ask you to quit.)
- 6. Compensation for study: If your health is harmed by participating in this study, our hospital will be responsible for providing treatment costs.
- 7. Confidentiality system: Your participation in this study will be confidential. The results will be published for scientific purposes without revealing your identity. Peking Union Medical College Hospital will keep all your records in this study as well as relevant hospital and office records.
- 8. Informed consent is in duplicate, one for each subject and one for the investigator, signed by both parties.

## Informed consent of subjects:

I have read and fully understood the above and have carefully considered the above, especially the rights, risks, and benefits of my participation in this study. I volunteered to participate in the study and was willing to cooperate with the investigator. At the same time, I declare that I can withdraw from this study at any time for any reason without losing any legal rights.

| Signature of Subject: | Date: |
|----------------------------|-------|
| Signature of Investigator: | Date: |